CLINICAL TRIAL: NCT01225419
Title: Mobilization by Plerixafor of Haematopoietic Stem Cells in Children
Acronym: MEP1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0082
Record Dates: First submitted 2010-10-05; First posted 2010-10-21 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Children Cancer, Solid Tumor
Keywords: Plerixafor; Hematopoietic Stem Cell Transplant mobilization; children
MeSH Terms: interventions — plerixafor

INTERVENTIONS:
Drug: Plerixafor, mozobil — Subcutaneous injection of 240 µg/kg of Plerixafor (Mozobil ®, Genzyme) at 8 am the day of the cytapheresis. Determination of CD34+ cells circulating in h0 then every hour of h3 to h11. Taking by cytapheresis from the 5th hour of the injection if the rate of CD34+ is upper or equal in 10.106/l. If the rate of CD34+ in the blood does not reach 10.106/l after the first injection of plerixafor or if the first cytapheresis does not allow the collection of at least 5.106/kg CD34+ cells, the patient will be considered in failure and a conventional mobilization by G-CSF will be programmed

SUMMARY:
This is a prospective Phase II, monocentre study.

DETAILED DESCRIPTION:
The extensive chemotherapy followed of hematopoietic stem cells reinjection (HSC) is one therapeutic option which the profit is well demonstrated in the treatment of children's solid tumors. It's one of the "standard" treatment of the following tumors: neuroblastoma, metastatic medulloblastoma, Ewing sarcoma, lymphoma in relapse; and because of the big chemosensibility of paediatric cancers, stays an important therapeutic option in the rhabdomyosarcoma in relapse or metastatic, nephroblastoma, etc. The stem cells can be taken in the blood by cytapheresis after mobilization with pharmacologic molecules. At present, the reference of the mobilization treatment is the G-CSF (Granulocyte colony-stimulating factor) in monotherapy during 4 to 6 days. His inconveniences are: lasted of the treatment (4 to 6 days), reproduction of the injections (1 to 2 subcutaneous injections daily), day variability of the peak of mobilization, this hematopoietic stimulation imposes to delay the chemotherapy. The plerixafor activates a massive and fast mobilization of the HSC ( hematopoietic stem cells)(between 6 and 11 hours after the injection). Currently, it's indicated in association with the G-CSF ( Granulocyte colony-stimulating factor)in case of mobilization failure. However, his big flexibility of use could be of a big interest in monotherapy at the child. To date, there is in our knowledge no data on the use of this molecule at the child.

Schema of study: Subcutaneous injection of 240 µg/kg of Plerixafor (Mozobil ®, Genzyme) at 8 am the day of the cytapheresis. Determination of CD34+ cells circulating in h0 then every hour of h3 to h11. Taking by cytapheresis from the 5th hour of the injection if the rate of CD34+ is upper or equal in 10.106/l. If the rate of CD34+ in the blood does not reach 10.106/l after the first injection of plerixafor or if the first cytapheresis does not allow the collection of at least 5.106/kg CD34+ cells, the patient will be considered in failure and a conventional mobilization by G-CSF(Granulocyte colony-stimulating factor) will be programmed.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 18 years old
* Solid malign tumor
* Lansky score ≥ 70%
* Indication of hematopoietic stem cell taking by cytapheresis for extensive chemotherapy followed by one or several reinjections of hematopoietic stem cells

Exclusion Criteria:

* Administration of hematopoietic growth factors in 8 days preceding the injection of Plerixafor.
* Contraindication in the cytapheresis or in the extensive chemotherapy.
* Clinical or biological state dissuading the realization of the cytapheresis
* Chemotherapy in 15 days preceding the injection of plerixafor or neutrophils < 1500/mm3

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Percentage of the children to whom 5.106 cells CD34 + / kg can be collected in 2 masses blood treated (one cytapheresis). | between H4 and H9 at day 0

SECONDARY OUTCOMES:
Describe the kinetics of mobilization of the hematopoietic progenitor at the child in situation of hematopoietic stable state after a subcutaneous injection of plerixafor | between the injection and the apheresis at day 0
Describe the pharmacokinetics of the plerixafor at the child | between the injection and the apheresis at day 0
Describe the side effects | day 0 to day 3
Describe the capacity of hematopoietic reconstruction of taken cells after mobilization by plerixafor only | during the 30 following days
the toxicity of the plerixafor at the child. | day 0 to day 3

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MERLIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France